

#### **Statistical Analysis Plan**

**Detailed Title:** A phase IV, randomised, open-label, controlled study to

assess the immunogenicity and safety of the diphtheria, tetanus, pertussis and inactivated poliovirus (DPT-IPV) vaccine Squarekids<sup>TM</sup> when co-administered with GSK Biologicals' oral live attenuated HRV liquid vaccine Rotarix<sup>TM</sup> in healthy Japanese infants aged 6 - 12 weeks at

the time of the first dose of HRV vaccination.

eTrack study number and Abbreviated Title

114720 (ROTA-079)

**Scope:** All data pertaining to the above study.

**SAP Version** Version 1

**SAP date** 12-SEP-2016

Co-ordinating author: PPD

Reviewed by: PPPClinical and Epidemiology Project Lead)

(Clinical Research and Development Lead)

PPD (Lead statistician)

(peer reviewer statistician),

PPD (Lead statistical analyst)

PPD (Scientific writer)

(Lead Scientific writer)

PPD (Regulatory Affair)

Proclinical Safety representative)

PP(CTRs)

**Approved by:** (Clinical and Epidemiology Project Lead)

delegating to PPD (Clinical Research and

Development Lead)

PPD (Lead statistician)

(Lead Scientific writer)

FORM-9000026972-01 Statistical Analysis Plan Template (Effective date: pilot for process, target to be effective in January 2017)

## **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| LIS | T OF A | ABBREVIATIONS | 6 |
| 1. | DOCUMENT HISTORY | | |
| 2. | STUD | Y DESIGN | 7 |
| 3. | OD IE | CTIVES | 0 |
| ა. | 3.1. | Primary objective | |
| | 3.2. | | |
| 4. | ENDF | POINTS | 10 |
| | 4.1. | Primary endpoint | |
| | 4.2. | Secondary endpoints | 10 |
| 5. | | YSIS SETS | |
| | 5.1. | Definition5.1.1. Total vaccinated cohort | |
| | | 5.1.2. According-to-protocol cohort for analysis of | |
| | | immunogenicity | 11 |
| | 5.2. | Criteria for eliminating data from Analysis Sets | |
| | | 5.2.1. Elimination from TVC | 12 |
| | | immunogenicity | 12 |
| | | 5.2.3. Right censored Data | 13 |
| | | 5.2.4. Visit-specific censored Data | |
| | 5.3. | Important protocol deviation not leading to elimination from per-<br>protocol analysis set | 13 |
| 6. | СТАТ | ISTICAL ANALYSES | 1.1 |
| 0. | 6.1. | Demography | |
| | 0.1. | 6.1.1. Analysis of demographics/baseline characteristics planned | |
| | | in the protocol | 14 |
| | | 6.1.2. Additional considerations | |
| | 6.2. | Exposure | 14 |
| | | 6.2.1. Analysis of exposure planned in the protocol | |
| | 6.3. | Immunogenicity | |
| | 0.0. | 6.3.1. Analysis of immunogenicity planned in the protocol | |
| | | 6.3.2. Additional considerations | 15 |
| | 6.4. | Analysis of safety | |
| | | 6.4.1. Analysis of safety planned in the protocol | |
| 7. | ANAL | YSIS INTERPRETATION | 18 |
| 8. | | | |
| Ο. | 8.1. | DUCT OF ANALYSESSequence of analyses | |
| | 8.2. | Statistical considerations for interim analyses | |

| 9. | CHAN | GES FRO | DM PLANNED ANALYSES | 114720 (ROTA-079)<br>Statistical Analysis Plan<br>19 |
|---|---|---|---|---|
| 10. | SPECI | IFICATIO | NS FOR TABLES, LISTINGS AND FIGURES | 19 |
| 11. | METH<br>11.1. | ODS<br>Statistic<br>Standard<br>11.2.1.<br>11.2.2.<br>11.2.3. | NDARD DATA DERIVATION RULE AND STATE al method references d data derivation Date derivation Dose number Demography Immunogenicity Safety Data presentation description | 20<br>20<br>20<br>20<br>20<br>21<br>21 |
| 12. | ANNE | X 2: SUM | IMARY ON ELIMINATION CODES | 24 |
| 13. | ANNE | X 3: STU | DY SPECIFIC MOCK TFL | 25 |

114720 (ROTA-079) Statistical Analysis Plan

## **LIST OF TABLES**

| | | PAGE |
|---------|-------------------------------------------------------|------|
| Table 1 | Study groups and epochs foreseen in the study | 7 |
| Table 2 | Study groups and treatment foreseen in the study | 8 |
| Table 3 | Sub-cohorts | 8 |
| Table 4 | Intervals between study visits for code 2080 and 2090 | 13 |

114720 (ROTA-079) Statistical Analysis Plan

## LIST OF FIGURES

| | | PAGE |
|----------|----------------------------------------------|------|
| Figure 1 | Sequence for evaluating the study objectives | 18 |

114720 (ROTA-079) Statistical Analysis Plan

#### LIST OF ABBREVIATIONS

AE Adverse event

ATP According-To-Protocol

CI Confidence Interval

BMI Body Mass Index

CTRS Clinical Trial Registry Summary

DPT Diphtheria, Pertussis and Tetanus toxoids

eCRF Electronic Case Report Form

ED50 Effective dose to inhibit 50% of the maximum

Eli Type Internal GSK database code for type of elimination code

FHA Filamentous Haemagglutinin

GMC Geometric mean antibody concentration

GMT Geometric mean antibody titer

GSK GlaxoSmithKline HRV Human Rotavirus IgA Immunoglobulin A

IPV Inactivated Poliovirus Vaccine IU/ml International unit per milliliter

LL Lower Limit of the confidence interval

LSLV Last Subject Last Visit

MedDRA Medical Dictionary for Regulatory Activities

PT Pertussis Toxoid

RV Rotavirus

SAE Serious adverse event SAP Statistical Analysis Plan

SBIR GSK Biological's Internet Randomization System

SD Standard Deviation

TFL Tables Figures and Listings

TOC Table of Content

TVC Total Vaccinated Cohort

UL Upper Limit of the confidence interval

U/ml Unit per milliliter

#### 1. DOCUMENT HISTORY

| Date | Description | Protocol Version |
|-------------|--------------------------|---------------------|
| 12-SEP-2016 | Version 1: first version | Final – 03-JUN-2016 |

### 2. STUDY DESIGN



N = Number of subjects planned to be enrolled; n = Number of subjects in each group; BS = Blood Sampling. Visit 3 and Visit 5 are applicable only for subjects in the Staggered group. Visit 4 is applicable only for subjects in the Co-administration group.

- Experimental design: Phase IV, open-label, randomised, controlled, multi-centric, single-country study with two parallel groups.
- Primary Completion Date: Visit 7 (Month 5)
- End of Study: Last testing results released of samples collected at Visit 7
- Study groups: The study groups and epoch foreseen in the study are provided in Table 1.

Table 1 Study groups and epochs foreseen in the study

| Study Groups | Number of aubicate | Ago (Min/ Mox) | Epoch |
|---|---|---|---|
| Study Groups | Number of subjects | Age (Min/ - Max) | Epoch 001 |
| Co-administration group | 146 | 6 weeks - 12 weeks | Х |
| Staggered group | 146 | 6 weeks - 12 weeks | Х |

• The study groups and treatment foreseen in the study are provided in Table 2.

Table 2 Study groups and treatment foreseen in the study

| Treatment name | Vaccine name | Study Groups | |
|----------------|--------------|-------------------------|-----------------|
| | | Co-administration group | Staggered group |
| Rotarix | HRV | X | X |
| Squarekids | Squarekids | X | X |

- Control: active control (Staggered group).
- Vaccination schedules: The vaccination schedules are as follows:
  - Subjects in the Co-administration group will be administered the DPT-IPV vaccine according to a 3, 4, 6 month schedule and the liquid HRV vaccine according to a 2, 3 month schedule.
  - Subjects in the Staggered group will be administered the DPT-IPV vaccine according to a 3, 4.5, 6 month schedule and the liquid HRV vaccine according to a 2, 3.5 month schedule.
- Treatment allocation: Randomised 1:1 using GSK Biologicals' central randomisation system on Internet (SBIR). The randomisation algorithm will use a minimisation procedure accounting for centre and stratified for a HRV immunogenicity subcohort.
- Blinding: Open-label.
- Sampling schedule: Details of the samples to be collected are as follows:
  - A blood sample of approximately 2 mL will be collected from a sub-cohort of subjects, 1 month after the administration of the second dose of the liquid HRV vaccine.
  - A blood sample of approximately 5 mL will be collected at Visit 7, 1 month after administration of the last dose of DPT-IPV vaccine from all the subjects.
- Details of the HRV Immunogenicity sub-cohort are provided in Table 3. The sub-cohort will consist of 146 subjects (the first 73 subjects enrolled into the study from each study group).

Table 3 Sub-cohorts

| Sub-cohort name | Description | Estimated number of |
|---|---|---|
| | | subjects |
| HRV Immunogenicity sub-cohort | The serum anti-RV IgA antibody concentration and seropositivity 1 month after the second dose of the liquid HRV vaccine will be assessed in this sub-cohort of subjects. | 146 subjects (approximately half the number of subjects (73) from each study group)* |

<sup>\*</sup> The first 73 subjects enrolled into each study group will be allocated to the sub-cohort.

• Recording of solicited local symptoms within 8 days follow-up period (Day 0 - Day 7) after the first dose of DPT-IPV vaccine.

- Recording of solicited general symptoms within 8 days follow-up period (Day 0 -Day 7) following administration of each dose of HRV vaccine and after the first dose of DPT-IPV vaccine.
- Recording of unsolicited symptoms within 31 days (Day 0- Day 30) following administration of each dose of HRV vaccine and after the first dose of DPT-IPV vaccine.
- Recording of causally related AEs from the first study vaccine up to Visit 7.
- Recording of SAEs from first study vaccine up to Visit 7.
- Recording of AEs/SAEs leading to withdrawal from the study from the first study vaccine.
- Recording of SAEs that are related to study participation (i.e. protocol-mandated procedures, invasive tests, a change from existing therapy) or are related to a concurrent GSK medication/vaccine from the time the subject consents to participate in the study until Visit 7.
- Type of study: self-contained.
- Data collection: Electronic Case Report Form (eCRF).

#### 3. OBJECTIVES

## 3.1. Primary objective

 To demonstrate that the immunogenicity to the antigens contained in DPT-IPV vaccine is not impaired by the co-administration with GSK Biologicals' liquid HRV vaccine.

Criteria for non-inferiority (1 month after the third dose of DPT-IPV vaccine at Visit 7):

- Lower limits of the standardised asymptotic 95% confidence intervals (CIs) on the differences (Co-administered group minus Staggered group) in the percentages of subjects with seroprotective concentrations ≥ 0.1 IU/mL for anti-diphtheria (anti-D) antibodies and concentrations ≥ 0.1 IU/mL for anti-tetanus (anti-T) antibodies are ≥-10% (clinical limit for non-inferiority),
- Lower limits of the 95% CIs on the differences (Co-administered group minus Staggered group) in the percentages of subjects with concentrations ≥ 10 IU/mL for antibodies against the pertussis toxoid (PT) and filamentous hemagglutinin (FHA) antigens (anti-PT and anti-FHA) are ≥ -10% (clinical limit for non-inferiority),
- Lower limits of the standardised asymptotic 95% CIs on the differences (Co-administered group minus Staggered group) in the percentages of subjects with seroprotective titres (≥8 ED<sub>50</sub>) for each of anti-poliovirus serotypes 1, 2 and 3 antibodies are  $\ge$  -10% (clinical limit for non-inferiority).

## 3.2. Secondary objectives

- To assess the immunogenicity of the liquid HRV vaccine in terms of serum anti-RV IgA antibody seropositivity and Geometric Mean Concentrations (GMCs) in a subcohort of subjects, 1 month after the second dose of the liquid HRV vaccine.
- To assess the immunogenicity to all the antigens contained in the DPT-IPV vaccine in terms of GMCs/ geometric mean antibody titres (GMTs), 1 month after the third dose of the DPT-IPV vaccine.
- To assess reactogenicity and safety after each dose of liquid HRV vaccine and first dose of DPT-IPV vaccine in terms of solicited symptoms during the 8-day follow-up period and unsolicited symptoms during the 31-day follow-up period.
- To assess safety in terms of serious adverse events (SAEs) from the first dose of study vaccine up to study end.

#### 4. ENDPOINTS

## 4.1. Primary endpoint

- Immunogenicity with respect to components of the DPT-IPV vaccine 1 month after administration of the third dose of the vaccine (Visit 7):
  - anti-diphtheria antibody concentrations  $\geq 0.1 \text{ IU/mL}$ ,
  - anti-tetanus antibody concentrations  $\geq 0.1 \text{ IU/mL}$ ,
  - anti-PT and anti-FHA antibody concentrations  $\geq 10 \text{ IU/mL}$ ,
  - anti-poliovirus serotypes 1, 2 and 3 antibody titre  $\geq$  8 ED<sub>50</sub>.

## 4.2. Secondary endpoints

- Serum anti-RV IgA antibody concentration and seropositivity in a sub-cohort of subjects, 1 month after the second dose of the liquid HRV vaccine.
- Serum GMCs/GMTs for anti-diphtheria, anti-tetanus, anti-poliovirus serotypes 1, 2 and 3, anti-PT and anti-FHA antibodies, 1 month after the third dose of the DPT-IPV vaccine.
- Occurrence of solicited general symptoms during the 8-day (Days 0-7) follow-up period after each dose of liquid HRV vaccine.
- Occurrence of solicited local and general symptoms during the 8-day (Days 0-7) follow-up period after the first dose of DPT-IPV vaccine.
- Occurrence of unsolicited AEs during the 31-day (Days 0-30) follow-up period after each dose of the liquid HRV vaccine and the first dose of DPT-IPV vaccine, according to the Medical Dictionary for Regulatory Activities (MedDRA) classification.
- Occurrence of SAEs from the first dose of the study vaccine up to study end (Visit 7).

#### 5. ANALYSIS SETS

#### 5.1. Definition

Two cohorts are defined for the purpose of the analysis:

- Total vaccinated cohort.
- ATP cohort for analysis of immunogenicity.

#### 5.1.1. Total vaccinated cohort

The TVC will include all subjects with at least one dose of the study vaccines administration documented:

- A safety and reactogenicity analysis based on the TVC will include all subjects with at least one vaccine administration documented.
- An immunogenicity analysis based on the TVC will include all subjects from this cohort for whom immunogenicity data were available.

The TVC analysis will be performed per treatment actually administered.

#### 5.1.2. According-to-protocol cohort for analysis of immunogenicity

The ATP cohort for immunogenicity will include all eligible subjects:

- who comply with vaccination schedule of DPT-IPV and HRV vaccines,
- for whom the DPT-IPV and HRV vaccines were administered according to protocol
- who have not received vaccine/medication forbidden by the protocol (up to Visit 7),
- whose underlying medical condition was not forbidden by the protocol (up to Visit 7),
- who complied with the blood sampling schedule at visit 7,
- who had no concomitant infection related to any component of the DPT-IPV vaccine which may have influenced the immune response up to blood sample at visit 7,
- who had no concomitant infection unrelated to any component of the DPT-IPV vaccine which may have influenced the immune response up to blood sample at visit 7. Note that RV GE will not be considered as concomitant infection unrelated to any component of the DPT-IPV vaccine.
- for whom immunogenicity data are available for at least one antigen of the DPT-IPV vaccine at visit 7 sampling time point.

## 5.2. Criteria for eliminating data from Analysis Sets

Elimination codes are used to identify subjects to be eliminated from analysis. Detail is provide below for each sets.

#### 5.2.1. Elimination from TVC

Code 1030 (Study vaccine dose not administered at all but subject number allocated) and code 900 (invalid informed consent or fraud data) will be used for identifying subjects eliminated from TVC.

## 5.2.2. Elimination from ATP cohort for analysis of immunogenicity

A subject will be excluded from the ATP cohort for analysis of immunogenicity under the following conditions:

| Code | Condition under which the code is used |
|---|---|
| Eli Type =MA | |
| 900 | Invalid informed consent or fraud data |
| 1030 | Study vaccine dose not administered at all but subject number allocated |
| 1040 | Administration of concomitant vaccine(s) forbidden in the protocol up to blood sample at visit 7 |
| 1050 | Randomisation failure (subject not randomized in the correct group) |
| 1070 | Study vaccine dose not administered according to protocol: |
| | - Site or route of study vaccine administration wrong or unknown |
| | - Administration not according to protocol for reason specified by the investigator other than site and route |
| | - Wrong replacement or study vaccine administered (not compatible with the vaccine regimen associated to the treatment number) |
| | - Only part of the multiple planned administrations at one visit has been administered |
| 1080 | Vaccine has been administered (effective treatment number) despite a temperature deviation qualified by Status QA GMP NON Use |
| 1090 | Vaccine has been administered (effective treatment number) out of the expiration date at the time of administration |
| 2010 | Protocol violation linked to the inclusion/exclusion criteria |
| 2040 | Administration of any medication forbidden by the protocol up to blood sample at visit 7 |
| 2050 | Underlying medical condition forbidden by the protocol up to blood sample at visit 7 |
| 2060 | Concomitant infection related to any component of the DPT-IPV vaccine which may influence the immune response up to blood sample at visit 7 |
| 2070 | Concomitant infection not related to any component of the DPT-IPV vaccine other than RV GE which may influence the immune response up to blood sample at visit 7. Note that RV GE will not be considered as concomitant infection unrelated to any component of the DPT-IPV vaccine. |
| 2080 | Non compliance with vaccination schedule for HRV and/or DPT-IPV vaccination – see Table 4 |
| 2090 | Non compliance with blood sample schedule at Visit 7 – see Table 4 |

| Code | Condition under which the code is used |
|---|---|
| Eli Type =MA | |
| 2100 | Essential serological data missing: serological data missing for all antigens in the DPT-IPV vaccine at Visit 7 |
| 2120 | Obvious incoherence, abnormal serology evolution or error in data (Eg; incoherence between CRF and results, wrong sample labelling) |

Table 4 Intervals between study visits for code 2080 and 2090

| Study Group | Interval | Optimal length of interval <sup>1</sup> | Allowed interval <sup>2</sup> |
|---|---|---|---|
| Co-administration group | Visit 1→Visit 2* | 30 days | 28 days - 42 days |
| | Visit 2→Visit 4 | 30 days | 28 days – 42days |
| | Visit 4→Visit 6 | 56 days | 28 days - 56 days |
| | Visit 6→Visit 7 | 30 days | 21 days - 48 days |
| Staggered group | Visit 1→Visit 2* | 30 days | 28 days - 42 days |
| | Visit 2→Visit 3 | 15 days | 7 days - 21 days |
| | Visit 3→Visit 5** | 30 days | 28 days - 42 days |
| | Visit 5→Visit 6 | 45 days | 28 days – 56 days |
| | Visit 6→Visit 7 | 30 days | 21 days - 48 days |

<sup>1.</sup> Whenever possible the investigator should arrange study visits within this interval.

There should be a time-period of at least 7 days between the administration of an inactivated vaccine and any other vaccine, and 28 days between the administration of a live virus vaccine and any other vaccine, in Japan. Please refer to the package inserts of *Rotarix* and *Squarekids* for more details.

#### 5.2.3. Right censored Data

Not applicable.

#### 5.2.4. Visit-specific censored Data

Not applicable.

# 5.3. Important protocol deviation not leading to elimination from per-protocol analysis set

The following important protocol deviations will be reported by groups:

• Forced randomization: in case of supplies shortage for the next assigned vaccine according to the randomization schedule at the clinical site, the randomization system will use the forced randomization procedure in order to continue to enrol and vaccinate subjects. The system moves seamlessly to the next treatment/randomization number for which vaccine supplies are available. The site will not be aware of the forced randomization event.

<sup>&</sup>lt;sup>2</sup>. Subjects will not be eligible for inclusion in the According To Protocol (ATP) cohort for analysis of immunogenicity if they make the study visit outside this interval.

<sup>\*</sup> Visit 2 should take place when the subject is 3 months of age or older.

<sup>\*\*</sup>The period between Visit 2 and Visit 5 should be within 8 weeks.

• Manual randomization: in case the randomization system is unavailable, the investigator has the option to perform randomization by selecting supplies available at the site according to a pre-defined rule.

#### 6. STATISTICAL ANALYSES

Note that standard data derivation rule and stat methods are described in Annex 1 and will not be repeated below.

#### 6.1. Demography

## 6.1.1. Analysis of demographics/baseline characteristics planned in the protocol

The distributions of subjects enrolled by centre will be tabulated by group.

The numbers of subjects who are withdrawn from the study will be tabulated by group according to the reason for withdrawal.

The median, mean, range and standard deviation (SD) of age at each study vaccine dose (in weeks) will be computed by group. The median, mean and SD of height in centimetre (cm) and weight in kilograms (kg) at Visit 1 will be computed by group. The Body Mass Index (BMI) at Visit 1 will also be computed as weight (in kg)/height<sup>2</sup> (in m). The gender composition per group will also be presented.

The deviations from specifications for age and intervals between study visits will be tabulated by group.

#### 6.1.2. Additional considerations

The median, mean, range and standard deviation (SD) of gestational age (in weeks) will be computed by group.

### 6.2. Exposure

#### 6.2.1. Analysis of exposure planned in the protocol

The number of doses of the liquid HRV vaccine and DPT-IPV vaccine administered will be tabulated per group.

#### 6.2.2. Additional considerations

None.

## 6.3. Immunogenicity

#### 6.3.1. Analysis of immunogenicity planned in the protocol

The ATP cohort for immunogenicity will be used for the primary analysis of immunogenicity. An analysis of immunogenicity based on the TVC will be performed

only if more than 5% of the vaccinated subjects with immunogenicity results available were excluded from the ATP cohort for immunogenicity. In such a case, the TVC analyses will evaluate whether exclusion from the ATP cohort has biased the results.

#### Within group assessment

For each treatment group and each antigen:

- Percentage of subjects with antibody concentrations/ titres greater than or equal to the pre-specified cut-off will be calculated with exact 95% CI (Refer Table 9 of the protocol). Anti-PT and anti-FHA antibody concentrations ≥ 10 IU/mL will also be calculated with exact 95% CI.
- GMC/GMTs, as applicable with 95% CIs will be computed.
- The distribution of antibody concentrations/ titres, as applicable, will be presented using reverse cumulative curves (RCCs).

#### Between group assessment

For each antigen in the DPT-IPV vaccine:

• The two-sided asymptotic standardised 95% CIs for the difference between groups (Co-administration group minus Staggered group) in terms of percentage of subjects with antibody concentrations/ titres greater than or equal to the pre-specified cut-off will be computed. Anti-PT and anti-FHA antibody concentrations ≥ 10 IU/mL will also be calculated with exact 95% CI.

#### 6.3.2. Additional considerations

The following seropositivity thresholds are applicable:

- anti-RV IgA antibody concentration  $\geq 20 \text{ U/mL}$ .
- anti- diphtheria antibody concentrations ≥ assay cut-off
- anti- tetanus antibody concentrations ≥ assay cut-off
- anti-PT antibody concentrations  $\geq 2.693 \text{ IU/mL}$
- anti-FHA antibody concentrations  $\geq 2.046 \text{ IU/mL}$

The following seroprotection thresholds are applicable:

- anti-diphtheria antibody concentrations  $\geq 0.1 \text{ IU/ml}$ ;
- anti-tetanus antibody concentrations ≥ 0.1 IU/ml;
- anti-poliovirus types 1, 2 and 3 antibody titres  $\geq 8$ .

Other cut-offs to be considered for summary tables and between-group comparisons

- Anti-PT antibody concentrations ≥ 10 IU/mL
- Anti-FHA antibody concentrations  $\geq 10 \text{ IU/mL}$

Anti-rotavirus IgA antibody GMCs and their 95% CI will also be computed on subjects seropositive for anti-rotavirus IgA antibody.

A sensitivity analysis excluding forced randomization will be performed for the primary objectives in case the percentage of forced randomizations exceed 5% (forced randomizations are allocation which were constrained by supply available at the site. In open studies, allocations without using the randomization system are also forced randomizations).

## 6.4. Analysis of safety

## 6.4.1. Analysis of safety planned in the protocol

The safety analysis will be based on the TVC.

The incidence by dose, overall per dose and overall per subject, with its exact 95% CI of

- any adverse event (solicited or unsolicited, local or general),
- at least one local adverse event (solicited or unsolicited), and,
- at least one general adverse event (solicited or unsolicited),

during the 8-day (Days 0-7) follow-up period will be tabulated. The same calculations will be performed for any Grade 3 (solicited or unsolicited) symptoms, related and for any adverse event requiring medical attention.

For each type of solicited symptom, the incidence during the 8-day (Days 0-7) follow-up period of the symptom (any grade, Grade 3, related, Grade 3 related, requiring medical advice) will be tabulated as follows:

- at each dose, the percentage of doses followed by the reporting of a symptom and its exact 95% CI.
- over all the doses, the percentage of subjects reporting the symptom and its exact 95% CI,
- over all the doses, the percentage of doses followed by the reporting of a symptom and its exact 95% CI.
- for fever, additional analyses will be performed by 0.5°C increments.

The percentage of subjects who receive concomitant medication, who receive antipyretic medication and prophylactic antipyretic medication during the 8-day (Days 0-7) and 31-day (Days 0-30) follow-up period post-vaccination will be tabulated by dose, overall per subject and over all the doses.

The verbatim reports of unsolicited symptoms will be reviewed by a physician and the signs and symptoms will be coded according to MedDRA. Every verbatim term will be matched with the appropriate Preferred Term. The percentage of subjects with unsolicited symptoms occurring during the 31 days (Days 0-30) with its exact 95% CI will be

114720 (ROTA-079) Statistical Analysis Plan

tabulated by preferred term. Similar tabulation will be done for Grade 3 unsolicited symptoms and for unsolicited symptoms causally related to vaccination.

Subjects who experienced at least one SAE during the entire study period (from the first dose till the end of the study [Visit 7]) will be reported and the SAEs will be described in detail.

#### 6.4.2. Additional considerations

- In line with the endpoint description separate analysis will be made for solicited symptom, unsolicited AE within 31 days post vaccination and concomitant medication for
  - o The 2 HRV doses
  - The first DTPa-IPV dose
- In line with the HRV project standard, the primary analysis of solicited symptom will be performed by administered dose regardless of whether a solicited symptom has been documented as present/absent. A complementary analysis by documented dose in which only dose for which presence/absence of the symptoms is recorded will performed in case the percentage of documented dose among administered dose exceed 5% for one visit or a group.
- The incidence by dose, overall per dose and overall per subject of any grade 3 adverse event (solicited or unsolicited, local or general) with causal relationship to vaccination during the 8-day (Days 0-7) follow-up period will be tabulated with exact 95% CI.
- The percentage of subjects with unsolicited symptoms requiring medical attention occurring within 31 days (Days 0-30) post-vaccination with its exact 95% CI will be tabulated by group and preferred term. Similar tabulation will also be done for unsolicited AEs rated as grade 3 in intensity with causal relationship to vaccination.
- The percentage of subjects with causally related AEs from the first study vaccine until Visit 7 will be tabulated by group and preferred term.
- Medications will be coded using the GSKDRUG dictionary. Medications which started during the specified periods (Days 0-7 and Days 0-30) will be counted rather than all medications taken during the specified periods.
- For clintrial.gov and EudraCT posting purposes, a summary of subjects with all
  combined solicited (regardless of their duration) and unsolicited adverse events will
  be provided. Solicited adverse events will be coded by MedDRA as per the
  following codes:

| Solicited symptom | Lower level code | Lower level term |
|----------------------------|------------------|---------------------------|
| Pain at injection site | 10022086 | Injection site pain |
| Redness at injection site | 10022098 | Injection site redness |
| Swelling at injection site | 10053425 | Injection site swelling |
| Fever | 10016558 | Fever |
| Irritability/Fussiness | 10057224 | Irritability postvaccinal |

| Solicited symptom | Lower level code | Lower level term |
|-------------------|------------------|------------------|
| Diarrhoea | 10012727 | Diarrhea |
| Vomiting | 10047700 | Vomiting |
| Loss of appetite | 10003028 | Appetite lost |
| Cough/ runny nose | 10011224 | Cough |
| Drowsiness | 10013649 | Drowsiness |

#### 7. ANALYSIS INTERPRETATION

Except for analysis on objectives with predefined success criterion and an appropriate type I error control (i.e. confirmatory analyses), no comparative analyses will be performed.

With respect to confirmatory analyses the interpretation must be done in a hierarchical manner.

Each objective can only be reached if the associated criteria is met and all previous objectives have been reached (see Figure 1).

Figure 1 Sequence for evaluating the study objectives



The sequence of testing for anti-poliovirus antibodies was based on the fact that polio type 2 is eradicated and serotype 1 is the most prevalent followed by type 3 as per a 10:1 ratio (cases confirmed worldwide in the calendar year 2012 [data in World Health Organization (WHO) headquarter as of 12 March 2013]).

#### 8. CONDUCT OF ANALYSES

## 8.1. Sequence of analyses

The final data analysis will include all data up to one month after the third dose of DPT-IPV vaccine. These analyses will include the final analysis of immunogenicity and the final analysis of solicited and unsolicited symptoms and SAEs from the first dose up to Visit 7.

| Description | Analysis<br>ID | Disclosure Purpose<br>(CTRS=web posting,<br>SR=study report,<br>internal) | Dry run review<br>needed (Y/N) | Study Headline<br>Summary (SHS)<br>requiring expedited<br>communication to<br>upper management<br>(Yes/No) | Reference for<br>TFL |
|---|---|---|---|---|---|
| Final<br>analysis | E1_01 | Study Report<br>CTRS | Y for in-text<br>tables, to be<br>generated<br>between<br>LSLV and 1<br>month<br>before Data<br>Base Freeze | Yes | All tables from<br>TFL dated<br>12-SEP-2016 |

## 8.2. Statistical considerations for interim analyses

All analyses will be conducted on final data and therefore no statistical adjustment for interim analyses is required.

#### 9. CHANGES FROM PLANNED ANALYSES

It was planned in the protocol to exclude subjects without any available results for both sampling time points (Visits 4/5 and 7) from the ATP cohort for analysis of immunogenicity. Actually, subjects without any available results for the sampling time point at Visit 7 will be excluded from the ATP cohort for analysis of immunogenicity.

# 10. SPECIFICATIONS FOR TABLES, LISTINGS AND FIGURES

The TFL TOC provides the list of tables/listings and figures needed for the study report. It also identifies the tables eligible for each analyses and their role (synopsis, in-text, post-text, SHS,...).

The following group names will be used in the TFLs:

| Group order in tables | Group label in tables | Group definition for footnote |
|---|---|---|
| 1 | Co-Administered | DPT-IPV vaccine administered according to a 3, 4, 6 month schedule and the liquid HRV vaccine according to a 2, 3 month schedule |
| 2 | Staggered | DPT-IPV vaccine administered according to a 3, 4.5, 6 month schedule and the liquid HRV vaccine according to a 2, 3.5 month schedule. |

# 11. ANNEX 1 STANDARD DATA DERIVATION RULE AND STATISTICAL METHODS

#### 11.1. Statistical method references

The exact two-sided 95% CIs for a proportion within a group will be the Clopper-Pearson exact CI [Clopper CJ, Pearson ES. The use of confidence or fiducial limits illustrated in the case of binomial. *Biometrika*. 1934;26:404-413].

The standardised asymptotic two-sided 95% CI for the group difference in proportions is based on the method described in the following paper:Robert G. Newcombe, interval estimation for the difference between independent proportions: comparison of eleven methods, *Statist Med.* 1998; 17, 873-890. The standardised asymptotic method used is the method six.

#### 11.2. Standard data derivation

#### 11.2.1. Date derivation

- SAS date derived from a character date: in case day is missing, 15 is used. In case day & month are missing, 30June is used.
- Onset day for an event (ae, medication, vaccination, ...): the onset day is the number of days between the last study vaccination & the onset/start date of the event. This is 0 for an event starting on the same day as a vaccination. See SAS date derived in case the start date of the event is incomplete.

#### 11.2.2. Dose number

- The study dose number is defined in reference to the number of study visits at which vaccination occurred. More specifically dose 1 refers to all vaccines administered at the first vaccination visit while dose 2 corresponds to all vaccinations administered at the second vaccination visit even if this is the first time a product is administered to the subject.
- Relative dose: the relative dose for an event (AE, medication, vaccination) is the most recent study dose given before an event. In case the event takes place on the day a study dose is given, the related dose will be that of the study dose, even if the event actually took place before vaccination. For instance, if an adverse event begins on the day of the study vaccination but prior to administration of the vaccine, it will be assigned to this dose. In case a study dose is not administered and an event occurs after the subsequent study dose (eg 3rd study dose), the relative dose of the event will be study dose associated to the subsequent study dose (eg dose 3).
- The number of doses for a product is the number of time the product was administered to a subject.
- The incidence per dose is the number of vaccination visits at which an event was reported among all vaccination visits.

#### 11.2.3. Demography

• Age: Age at the reference activity, computed as the number of units between the date of birth and the reference activity.

#### 11.2.4. Immunogenicity

- For a given subject and given immunogenicity measurement, missing or non-evaluable measurements will not be replaced.
- The Geometric Mean Concentrations/Titres (GMC/Ts) calculations are performed by taking the anti-log of the mean of the log titre transformations. Antibody titres below the cut-off of the assay will be given an arbitrary value of half the cut-off of the assay for the purpose of GMT calculation. The cut-off value is defined by the laboratory before the analysis and is described in Section 5.7.3 of the protocol.
- A seronegative subject is a subject whose antibody titre is below the cut-off value of the assay. A seropositive subject is a subject whose antibody titre is greater than or equal to the cut-off value of the assay.
- A seroprotected subject is a subject whose antibody concentration/titre is greater than or equal to the level defining clinical protection.
- The assay cut-off is the value under which there is no quantifiable result available. For an assay with a specific 'cut\_off', numerical immuno result is derived from a character field (rawres):
  - If rawres is 'NEG' or '-' or '(-)', numeric result= cutt\_off/2,
  - if rawres is 'POS' or '+' or '(+)', numeric result = cut off,
  - if rawres is '< value' and value<=cut off, numeric result =cut off/2,
  - if rawres is '< value' and value>cut off, numeric result =value,
  - if rawres is '> value' and value<cut off, numeric result =cut off/2,
  - if rawres is '> value' and value>=cut off, numeric result =value,
  - if rawres is '<= value' or '>= value' and value<cut\_off, numeric result =cut\_off/2.</p>
  - if rawres is '<= value' or '>= value' and value>=cut off, numeric result =value,
  - if rawres is a value < cut off, numeric result = cut off/2,
  - if rawres is a value >= cut off, numeric result = rawres,
  - if rawres is a value >= cut off. numeric result = rawres.
  - else numeric result is left blank.
- All CI computed will be two-sided 95% CI.

#### 11.2.5. Safety

• For analysis of solicited, unsolicited adverse events (such as serious adverse events or adverse events by primary MedDRA term) and for the analysis of concomitant medications, all vaccinated subjects will be considered. Subjects who did not report the event or the concomitant medication will be considered as subjects without the event or the concomitant medication respectively.

114720 (ROTA-079) Statistical Analysis Plan

- In case there will be more than 5% of subjects without documented dose for solicited symptoms (i.e., symptom screen not completed), sensitivity analysis will include only vaccinated subjects for doses with documented safety data (i.e., symptom screen completed).
- The following rules will be used for the analysis of solicited symptoms:
  - Subject who didn't document the presence or absence of a solicited symptom
    after one dose will be considered not having that symptom after that dose in the
    analysis done on "administrated dose"
  - Subjects who documented the absence of a solicited symptom after one dose will be considered not having that symptom after that dose.
  - Subjects who documented the presence of a solicited symptom and fully or
    partially recorded daily measurement over the solicited period will be included in
    the summaries at that dose and classified according to their maximum observed
    daily recording over the solicited period.
  - Subjects who documented the presence of a solicited symptom after one dose without having recorded any daily measurement will be considered as having that symptom after that dose).
- The maximum intensity of local injection site redness/swelling will be coded as follows:

| Grade | Redness/swelling |
|-------|--------------------|
| 0 | Absent |
| 1 | > 0 mm and ≤ 5 mm |
| 2 | > 5 mm and ≤ 20 mm |
| 3 | > 20 mm |

• For the analysis, temperatures will be coded as follows for oral, axillary or tympanic route:

| Grade | Temperature |
|-------|---------------------|
| 0 | < 37.5°C |
| 1 | ≥ 37.5°C - ≤ 38.0°C |
| 2 | > 38.0°C - ≤ 39.0°C |
| 3 | > 39.0°C |

For rectal route, temperatures will be converted to axillary setting by subtracting  $0.5^{\circ}$ 

• Note that for all tables described in this section, the way the percentage of subjects will be derived will depend on the event analysed (see table below for details). As a result, the N value will differ from one table to another.

114720 (ROTA-079) Statistical Analysis Plan

| Event | N used for deriving % per subject for<br>Vaccination phase | N used for deriving % per dose for Vaccination phase |
|---|---|---|
| Concomitant vaccination | All subjects with study vaccine administered | All study visits with study vaccine administered |
| Solicited general symptom | Primary analysis: all subjects with study vaccine administered | Primary analysis: all study visits with study vaccine administered |
| | Sensitivity analysis: all subjects with at least one solicited general symptom documented as either present or absent (i.e., symptom screen completed) | Sensitivity analysis: all study visits with study vaccine administered and with at least one solicited general symptom documented as either present or absent (i.e., symptom screen completed) |
| Solicited local symptom | Primary analysis: all subjects with study vaccine administered | Primary analysis: all study visits with study vaccine administered |
| | Sensitivity analysis: all subjects with at least one solicited local symptom documented as either present or absent (i.e., symptom screen completed) | Sensitivity analysis: all study visits with study vaccine administered and with at least one solicited local symptom documented as either present or absent (i.e., symptom screen completed) |
| Unsolicited symptom | All subjects with study vaccine administered | All study visits with study vaccine administered |
| Concomitant medication | All subjects with study vaccine administered | All study visits with study vaccine administered |

• All CI computed will be two-sided 95% CI.

## 11.2.6. Data presentation description

The following decimal description from the decision rules will be used for the demography, immunogenicity and safety/reactogenicity.

| Display Table | Parameters | Number of decimal digits |
|---|---|---|
| All summaries | % of count, including LL & UL of CI | 1 |
| Demographic characteristics | Mean, median, SD | 1 |
| Immunogenicity | % of difference, including LL & UL of CI | 2 |
| Immunogenicity | Anti-RV IgA GMC | 1 |
| Immunogenicity | Anti-diphtheria and anti-tetanus GMC | 1 |
| Immunogenicity | Anti-poliovirus serotypes 1, 2 and 3 GMT | 1 |
| Immunogenicity | Anti-PT and anti-FHA GMC | 1 |

## 12. ANNEX 2: SUMMARY ON ELIMINATION CODES

Refer to Section 5.2.

#### 13. ANNEX 3: STUDY SPECIFIC MOCK TFL

The following draft study specific mock will be used. The data display, title and footnote are for illustration purpose and will be adapted to the study specificity as indicated in the TFL TOC. These templates were copied from ROTA-056, Study Report/DTPa-HBV-IPV-125 and additional web tables were added. Note that there may be few changes between the study specific SAP mock TFL and the final TFLs. These editorial/minor changes will not lead to a SAP amendment.

| Template 1 | Number of subjects by centre (Total vaccinated cohort) | 28 |
|---|---|---|
| Template 2 | Number of subjects vaccinated, completed and withdrawn with reason for withdrawal at Visit 4 – First year conclusion (Total vaccinated cohort) | 28 |
| Template 3 | Number of subjects at each visit and list of withdrawn subjects up to visit 4 – First year conclusion (Total vaccinated cohort) | 29 |
| Template 4 | Number of subjects in the sub-cohorts (Total vaccinated cohort) | 29 |
| Template 5 | Number of subjects enrolled into the study as well as the number excluded from ATP analyses (Reactogenicity/Safety and Immunogenicity) with reasons for exclusion | 30 |
| Template 6 | Summary of demographic characteristics (ATP cohort for Immunogenicity) | 31 |
| Template 7 | Minimum and maximum activity dates (Total vaccinated cohort) | 32 |
| Template 8 | Deviations from specifications for age and intervals between study visits (Total vaccinated cohort) | 33 |
| Template 9 | Study population (Total vaccinated cohort) | 33 |
| Template 10 | Anti-rotavirus IgA antibody GMC and seropositivity rates - ATP cohort for immunogenicity | 34 |
| Template 11 | Anti-rotavirus IgA antibody GMC calculated on subjects seropositive for anti-rotavirus IgA antibodies - ATP cohort for immunogenicity | 34 |
| Template 12 | Seroprotection rates and GMC for anti-Diphtheria and anti-<br>Tetanus antibody concentrations by groups at pre booster<br>vaccination (ATP cohort for analysis of antibody persistence) | 34 |
| Template 13 | Seropositivity rates and GMC for anti-PT by groups at pre booster vaccination (ATP cohort for analysis of antibody persistence) | 35 |
| Template 14 | Seroprotection rates and geometric mean titres (GMT) for anti-<br>Poliovirus 1, 2 and 3 antibody by groups at pre vaccination (ATP cohort for analysis of antibody persistence) | 35 |

114720 (ROTA-079) Statistical Analysis Plan

| Template 15 I | Difference between groups in percentage of subjects with titre/concentrations equal to or above the proposed cut-off one month after primary vaccination between Form A and Control | |
|---|---|---|
| | groups - Inferential analysis (ATP cohort for immunogenicity) | 36 |
| Template 16 | Reverse Cumulative curves for anti-rotavirus IgA antibody concentrations at Visit 3 from a subset of subjects - ATP cohort for immunogenicity | 37 |
| Template 17 | Number and percentage of subjects who received study vaccine doses by vaccine (Total vaccinated cohort) | 38 |
| Template 18 | Compliance in returning symptom sheets (Total vaccinated cohort) | 38 |
| Template 19 | Incidence and nature of symptoms (solicited and unsolicited) reported during the 8-day (Days 0-7) post-vaccination period following each dose and overall (Total vaccinated cohort) | 39 |
| Template 20 | Incidence of solicited local symptoms reported during the 7-day (Days 0-6) post-vaccination period following each dose and overall (Total vaccinated cohort) | 39 |
| Template 21 | Incidence of solicited general symptoms reported during the 7-day (Days 0-6) post-vaccination period following each dose and overall (Total vaccinated cohort) | 40 |
| Template 22 | Incidence of solicited local symptoms reported during the 7-day (Days 0-6) post-vaccination period following each dose and overall (Total vaccinated cohort) | 42 |
| Template 23 | Incidence of solicited general symptoms reported during the 7-day (Days 0-6) post-vaccination period following each dose and overall (Total vaccinated cohort) | 43 |
| Template 24 | Percentage of subjects reporting the occurrence of unsolicited symptoms classified by MedDRA Primary System Organ Class within the 31-day (Days 0-30) post-vaccination period (Total vaccinated cohort) | 45 |
| Template 25 | Percentage of doses with unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term within the 43-day (Days 0-42) post-vaccination period (Total vaccinated cohort) | 45 |
| Template 26 I | isting of dropouts due to AEs, SAEs and solicited symptoms (Total cohort) | 46 |
| Template 27 | Listings of SAEs (Total vaccinated cohort) | 47 |
| Template 28 | Number and percentage of doses and of subjects who took at least one concomitant medication during the study period (from Dose 1 till database lock) by type (Total vaccinated cohort) | 48 |
| | bood i illi databado look, by typo ( rotal vaccillated collect, | |

114720 (ROTA-079) Statistical Analysis Plan

| | Statistical Analysis | i iaii |
|---|---|---|
| Template 29 | Incidence of solicited general symptoms reported during the 7-day (Days 0-6) post-vaccination period following each dose and overall (Total vaccinated cohort) | 49 |
| Template 30 | Number (%) of subjects with serious adverse events from first study vaccination up to Visit 7 including number of events reported (Total vaccinated cohort) | 50 |
| Template 31 S | Solicited and unsolicited symptoms experienced by at least 5 % of subjects classified by MedDRA Primary System Organ Class and Preferred Term within 31-day (Days 0-30) post-vaccination period after any dose of liquid HRV vaccine and first dose of DPT-IPV vaccine - SAE excluded (Total vaccinated cohort) | 50 |
| Template 32 | Number of enrolled subjects by age category (Total vaccinated cohort) | 51 |

Template 1 Number of subjects by centre (Total vaccinated cohort)

| | HRV | Placebo | Tot | al |
|--------|-----|---------|-----|------|
| Center | n | n | n | % |
| PPD | 26 | 14 | 40 | 5.2 |
| PPD | 28 | 14 | 42 | 5.5 |
| PPD | 18 | 8 | 26 | 3.4 |
| PPD | 26 | 13 | 39 | 5.1 |
| PPD | 18 | 10 | 28 | 3.7 |
| PPD | 12 | 7 | 19 | 2.5 |
| PPD | 13 | 7 | 20 | 2.6 |
| PPD | 38 | 19 | 57 | 7.5 |
| PPD | 13 | 7 | 20 | 2.6 |
| PPD | 68 | 34 | 102 | 13.3 |
| PPD | 32 | 16 | 48 | 6.3 |
| PPD | 14 | 7 | 21 | 2.7 |
| PPD | 16 | 8 | 24 | 3.1 |
| PPD | 6 | 4 | 10 | 1.3 |
| PPD | 48 | 24 | 72 | 9.4 |
| PPD | 48 | 24 | 72 | 9.4 |
| PPD | 72 | 35 | 107 | 14.0 |
| PPD | 3 | 2 | 5 | 0.7 |
| PPD | 3 | 2 | 5 | 0.7 |
| PPD | 6 | 2 | 8 | 1.0 |
| All | 508 | 257 | 765 | 100 |

n = number of subjects included in each group or in total for a given centre or for all centres

All = sum of all subjects in each group or in total (sum of all groups)

 $% = n/AII \times 100$ 

Centre = GSK Biologicals' assigned centre number

Template 2 Number of subjects vaccinated, completed and withdrawn with reason for withdrawal at Visit 4 – First year conclusion (Total vaccinated cohort)

| | HRV | Placebo | Total |
|---|---|---|---|
| Number of subjects vaccinated | 508 | 257 | 765 |
| Number of subjects completed | 492 | 247 | 739 |
| Number of subjects withdrawn | 16 | 10 | 26 |
| Reasons for withdrawal: | | | |
| Serious Adverse Event | 1 | 0 | 1 |
| Non-serious adverse event | 0 | 1 | 1 |
| Protocol violation | 0 | 1 | 1 |
| Consent withdrawal (not due to an adverse event) | 9 | 3 | 12 |
| Migrated/moved from study area | 6 | 2 | 8 |
| Lost to follow-up (subjects with incomplete vaccination course) | 0 | 0 | 0 |
| Lost to follow-up (subjects with complete vaccination course) | 0 | 3 | 3 |
| Other - not reached | | | |
| Other - practical difficulty this year | | | |

Vaccinated = number of subjects who were vaccinated in the study

Completed = number of subjects who completed Visit 4

Withdrawn = number of subjects who did not come for Visit 4

Template 3 Number of subjects at each visit and list of withdrawn subjects up to visit 4 – First year conclusion (Total vaccinated cohort)

| Group | VISIT | N | Withdrawn<br>Subject numbers | Reason for withdrawal |
|---|---|---|---|---|
| HRV | VISIT 1 | 508 | | |
| | | | no. PP | CONSENT WITHDRAWAL |
| | | | no. PP | CONSENT WITHDRAWAL |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | VISIT 2 | 504 | | |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | | | no. PPD | SERIOUS ADVERSE EXPERIENCE |
| | VISIT 3 | 501 | | |
| | | | no | MIGRATION FROM STUDY AREA |
| | | | no. PP | CONSENT WITHDRAWAL |
| | | | no. PP | MIGRATION FROM STUDY AREA |
| | | | no. PP | CONSENT WITHDRAWAL |
| | | | no. PP | MIGRATION FROM STUDY AREA |
| | | | no. PP | MIGRATION FROM STUDY AREA |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | | | no. PPD | MIGRATION FROM STUDY AREA |
| | | | no. PPD | MIGRATION FROM STUDY AREA |
| | VISIT 4 | 492 | | |
| Placebo | VISIT 1 | 257 | | |
| | | | no. PP | PROTOCOL VIOLATION |
| | | | no. PP | CONSENT WITHDRAWAL |
| | VISIT 2 | 255 | | |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | VISIT 3 | 254 | | |
| | | | no. PP | MIGRATION FROM STUDY AREA |
| | | | no. PP | LOST TO FOLLOW-UP |
| | | | no. PP | LOST TO FOLLOW-UP |
| | | | no. PP | CONSENT WITHDRAWAL |
| | | | no. PP | MIGRATION FROM STUDY AREA |
| | | | no. PPD | LOST TO FOLLOW-UP |
| | | | no. PPD | ADVERSE EXPERIENCE |
| | VISIT 4 | 247 | | |

Template 4 Number of subjects in the sub-cohorts (Total vaccinated cohort)

| | | HF<br>N = 1 | | Placeb<br>N = 166 | - | Total<br>N = 3333 | |
|---|---|---|---|---|---|---|---|
| Characteristics | Categories | n | % | n | % | n | % |
| Sub-cohort | Immunogenicity sub cohort 1 | 306 | 18.4 | 306 | 18.4 | 612 | 18.4 |
| | Immunogenicity sub cohort 2 | 153 | 9.2 | 153 | 9.2 | 306 | 9.2 |

N = number of subject number

n = number of subject number in a given category

% = n / Number of subject number with available results x 100

114720 (ROTA-079) Statistical Analysis Plan

Template 5 Number of subjects enrolled into the study as well as the number excluded from ATP analyses (Reactogenicity/Safety and Immunogenicity) with reasons for exclusion

| | | Total | | H | RV | Placebo | |
|---|---|---|---|---|---|---|---|
| Title | n | S | % | n | S | n | S |
| Total cohort | 765 | | | | | | |
| Total vaccinated cohort | 765 | | 100 | 508 | | 257 | |
| Randomisation code broken at the investigator site ( code 1060 ) | 1 | 1 | | 1 | 1 | 0 | 0 |
| Essential serological data missing ( code 2100 ) | 3 | 3 | | 3 | 3 | 0 | 0 |
| Subject not planned to be bled for their all blood sampling visits ( code 2130 ) | 707 | 708 | | 470 | 471 | 237 | 237 |
| ATP cohort for immunogenicity | 54 | | 7.1 | 34 | | 20 | |

Note: Subjects may have more than one elimination code assigned

n = number of subjects with the elimination code assigned excluding subjects who have been assigned a lower elimination code number

s = number of subjects with the elimination code assigned

<sup>% =</sup> percentage of subjects in the considered ATP cohort relative to the Total vaccinated cohort

Template 6 Summary of demographic characteristics (ATP cohort for Immunogenicity)

| | | HF<br>N = | | Plac<br>N = | | To: | |
|---|---|---|---|---|---|---|---|
| | | Value or | % | Value or | % | Value or | % |
| Characteristics | Parameters or Categories | n | | n | | n | |
| Age (weeks) at Dose 1 of | | 7.5 | - | 7.2 | - | 7.4 | - |
| HRV | SD | 1.60 | - | 1.23 | - | 1.47 | - |
| | Median | 7.0 | - | 7.0 | - | 7.0 | - |
| | Minimum | 6 | - | 6 | - | 6 | - |
| | Maximum | 12 | - | 10 | - | 12 | - |
| Age (weeks) at Dose 2 of | Mean | 12.7 | - | 12.0 | - | 12.4 | - |
| HRV | SD | 1.57 | - | 1.45 | - | 1.55 | - |
| | Median | 12.0 | - | 12.0 | - | 12.0 | - |
| | Minimum | 11 | - | 10 | - | 10 | - |
| | Maximum | 11 | _ | 10 | - | 10 | - |
| | Missing | 17 | _ | 15 | - | 17 | - |
| Age (weeks) at Dose 1 of | | 12.7 | - | 12.0 | - | 12.4 | - |
| DPT-IPV | SD | 1.57 | - | 1.45 | - | 1.55 | - |
| 21 1 II V | Median | 12.0 | _ | 12.0 | - | 12.0 | _ |
| | Minimum | 11 | _ | 10 | _ | 10 | _ |
| | Maximum | 11 | _ | 10 | - | 10 | _ |
| | Missing | 17 | _ | 15 | _ | 17 | |
| Age (weeks) at Dose 2 of | | 17 | | 10 | | 17 | |
| DPT-IPV | SD | | | | | | |
| טו ו-וו ע | Median | | | | | | |
| | Minimum | | | | | | |
| | Maximum | | | | | | |
| | Missing | | | | | | |
| Ago (wooks) at Doos 2 of | | | | | | | |
| Age (weeks) at Dose 3 of DPT-IPV | SD | | | | | | |
| DP1-IPV | | | | | | | |
| | Median | | | | | | |
| | Minimum | | | | | | |
| | Maximum | | | | | | |
| | Missing | | 44.0 | | 70.0 | | -10 |
| Gender | Female | 14 | 41.2 | 14 | 70.0 | 28 | 51.9 |
| | Male | 20 | 58.8 | 6 | 30.0 | 26 | 48.1 |
| Geographical ancestry | African heritage / African | 0 | - | 0 | - | 0 | - |
| | American | | | _ | | _ | |
| | American Indian or Alaskan | 0 | - | 0 | - | 0 | - |
| | native | | | | | | |
| | Asian - Central/South Asian | 0 | - | 0 | - | 0 | - |
| | heritage | • | | _ | | _ | |
| | Asian - East Asian heritage | 0 | - | 0 | - | 0 | - |
| | Asian - Japanese heritage | 34 | 100 | 20 | 100 | 54 | 100 |
| | Asian - South east Asian | 0 | - | 0 | - | 0 | - |
| | heritage | • | | | | | |
| | Native Hawaiian or other Pacific Islande | 0 | | 0 | | 0 | |
| | White - Arabic / North African heritage | 0 | - | 0 | - | 0 | - |
| | White - Caucasian / European | 0 | - | 0 | - | 0 | - |
| | heritage | 0 | | _ | | | |
| | Other | 0 | - | 0 | - | 0 | - |

114720 (ROTA-079) Statistical Analysis Plan

| | | HR<br>N = 1 | Place<br>N = 1 | | Total<br>N = 54 | | |
|---|---|---|---|---|---|---|---|
| | | Value or | % | Value or | % | Value or | % |
| Characteristics | Parameters or | n | | n | | n | |
| | Categories | | | | | | |
| Height (cm) at visit 1 | Mean | 55.3 | - | 55.7 | - | 55.5 | - |
| | SD | 3.80 | - | 1.87 | - | 3.21 | - |
| | Median | 55.5 | - | 55.0 | - | 55.0 | - |
| Weight (kg) at visit 1 | Mean | 5.2 | - | 5.1 | - | 5.1 | - |
| J ( J, | SD | 0.66 | - | 0.49 | - | 0.60 | - |
| | Median | 5.1 | - | 5.2 | - | 5.2 | - |
| BMI at visit 1 (kg/m²) | Mean | | | | | | |
| , | SD | | | | | | |
| | Median | | | | | | |
| Gestational age (weeks) | Mean | | | | | | |
| , | SD | | | | | | |
| | Median | | | | | | |
| | Minimum | | | | | | |
| | Maximum | | | | | | |

N = total number of subjects in each group n = number of subjects in a given category

Value = value of the considered parameter % = n / Number of subjects with available results x 100

SD= standard deviation

Database Lock Date = 31MAR2009

## Template 7 Minimum and maximum activity dates (Total vaccinated cohort)

| Visit | Minimum date | Maximum date |
|-------|--------------|--------------|
| 1 | 19JUN2007 | 29DEC2007 |
| 2 | 24JUL2007 | 08FEB2008 |
| 3 | 24AUG2007 | 18MAR2008 |
| 4 | 25MAR2008 | 22NOV2008 |
| 5 | 24MAR2009 | 31MAR2009* |

<sup>\*</sup>Database Lock Date = 31MAR2009

Template 8 Deviations from specifications for age and intervals between study visits (Total vaccinated cohort)

| | | Age | PRE-Dose:1 | Dose:1 | -Dose:2 | Dose:2 | -PII(M2) |
|---|---|---|---|---|---|---|---|
| Group | | Protocol | Protocol | Protocol | Adapted | Protocol | Adapted |
| | | from 6 to 14 weeks | from 0 to 0 days | from 30 to | from 21 to | from 30 to | from 21 to |
| | | | | 48 days | 48 days | 48 days | 48 days |
| HRV | N | 508 | 37 | 499 | 499 | 35 | 35 |
| | n | 0 | 0 | 0 | 0 | 0 | 0 |
| | % | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 |
| | range | 6 to 14 | 0 to 0 | 30 to 47 | 30 to 47 | 30 to 45 | 30 to 45 |
| Placebo | N | 257 | 20 | 250 | 250 | 20 | 20 |
| | n | 1 | 0 | 0 | 0 | 0 | 0 |
| | % | 0.4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 |
| | range | 5 to 14 | 0 to 0 | 30 to 47 | 30 to 47 | 30 to 42 | 30 to 42 |

Adapted = interval used for defining the ATP cohorts for immunogenicity

N = total number of subjects with available results

n (%) = number / percentage of subjects with results outside of the interval

range = minimum-maximum for age and intervals

PRE = pre-vaccination

PII(M2) = One month after the second dose (Visit 3)

Template 9 Study population (Total vaccinated cohort)

| Number of subjects | [each group] | Total |
|---|---|---|
| Planned, N | | |
| Randomised, N ( <total cohort="" vaccinated="">)</total> | | |
| Completed, n (%) | | |
| Demographics | | |
| N ( <total cohort="" vaccinated="">)</total> | | |
| Females:Males | | |
| Mean Age, <years> (SD)</years> | | |
| Median Age, <years> (minimum, maximum)</years> | | |
| <most category="" frequent="" of="" race="">, n (%)</most> | | |
| <second category="" frequent="" most="" of="" race="">, n (%)</second> | | |
| <third category="" frequent="" most="" of="" race="">, n (%)</third> | | |

[each group]:

Short group label= long group label

## Template 10 Anti-rotavirus IgA antibody GMC and seropositivity rates - ATP cohort for immunogenicity

| | | | | ≥ 20 l | J/mL | | | GMC | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95% CI | | | 95% | 6 CI |
| Group | Timing | N | n | % | LL | UL | value | LL | UL |
| HRV | PRE | 34 | 0 | 0.0 | 0.0 | 10.3 | <20 | - | - |
| | PII(M2) | 34 | 29 | 85.3 | 68.9 | 95.0 | 217.0 | 109.9 | 428.6 |
| Placebo | PRE | 20 | 0 | 0.0 | 0.0 | 16.8 | <20 | - | - |
| | PII(M2) | 20 | 1 | 1 5.0 | | 24.9 | <20 | <20 - | |

GMC = geometric mean antibody concentration calculated on all subjects

N = number of subjects with available results

n (%) = number (percentage) of subjects with concentration ≥ 20 U/mL

95% CI = 95% confidence interval; LL = Lower Limit, UL = Upper Limit

PII (M2) = One month after the second dose (Visit 3)

PRE = pre-vaccination

Template 11 Anti-rotavirus IgA antibody GMC calculated on subjects seropositive for anti-rotavirus IgA antibodies - ATP cohort for immunogenicity

| | | | GMC | | |
|---------|---------|----|-------|-------|-------|
| | | | | 95% | CI |
| Group | Timing | N | value | LL | UL |
| HRV | PII(M2) | 29 | 368.9 | 202.1 | 673.3 |
| Placebo | PII(M2) | 1 | 496.0 | - | - |

GMC = geometric mean antibody concentration calculated on subjects with concentration ≥ 20 U/mL

N = number of subjects who seroconverted for Anti-rotavirus IgA Antibody

95% CI = 95% confidence interval; LL = Lower Limit, UL = Upper Limit

PII (M2) = One month after the second dose (Visit 3)

Template 12 Seroprotection rates and GMC for anti-Diphtheria and anti-Tetanus antibody concentrations by groups at pre booster vaccination (ATP cohort for analysis of antibody persistence)

| | | | | ≥ 0.1 IU/ml | | | | | ≥1 | IU/m | l | GMC | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | 95% CI | | :1 | | 95% CI | | | 95% | 6 CI |
| Antibody | Group | Timing | N | n | % | LL | UL | n | % | LL | UL | value | LL | UL |
| Anti- Diphtheria | Group A | Pre-BST | 271 | 241 | 88.9 | 84.6 | 92.4 | 1 | 0.4 | 0.0 | 2.0 | 0.175 | 0.163 | 0.188 |
| · | Group B | Pre-BST | 272 | 250 | 91.9 | 88.0 | 94.9 | 0 | 0.0 | 0.0 | 1.3 | 0.189 | 0.176 | 0.202 |
| | Control | Pre-BST | 279 | 234 | 83.9 | 79.0 | 88.0 | 2 | 0.7 | 0.1 | 2.6 | 0.154 | 0.142 | 0.166 |
| Anti-Tetanus | Group A | Pre-BST | 272 | 269 | 98.9 | 96.8 | 99.8 | 8 | 2.9 | 1.3 | 5.7 | 0.450 | 0.423 | 0.478 |
| | Group B | Pre-BST | 273 | 271 | 99.3 | 97.4 | 99.9 | 10 | 3.7 | 1.8 | 6.6 | 0.509 | 0.481 | 0.540 |
| | Control | Pre-BST | 278 | 275 | 98.9 | 96.9 | 99.8 | 6 | 2.2 | 0.8 | 4.6 | 0.380 | 0.359 | 0.404 |

Group A = Subjects who received DTPa-IPV/Hib vaccine at 2, 3, 4 months of age in the primary study

Group B = Subjects who received DTPa-IPV/Hib vaccine at 3, 4, 5 months of age in the primary study

Control = Subjects who received DTPa/Hib + IPV vaccines at 2, 3, 4 months of age in the primary study

Seroprotection=Anti-Diphtheria and Anti-Tetanus antibody concentration ≥0.1 IU/ml

GMC = geometric mean antibody concentration calculated on all subjects

N = number of subjects with available results

n/% = number/percentage of subjects with concentration equal to or above specified value

95% CI = 95% confidence interval; LL = Lower Limit, UL = Upper Limit

Pre-BST=Pre-booster vaccination blood sampling time point

## Template 13 Seropositivity rates and GMC for anti-PT by groups at pre booster vaccination (ATP cohort for analysis of antibody persistence)

| | | | | | ≥ 2.693 IU/mL | | | | | ≥ 10 IU/mL | | | | GMC |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95% CI | | | | 95% CI | | | | 95% ( | |
| Antibody | Group | Timing | N | n | % | LL | UL | n | % | LL | UL | value | LL | UL |
| Anti-PT | Group A | Pre-BST | 272 | 260 | 95.6 | 92.4 | 97.7 | 38 | 14.0 | 10.1 | 18.7 | 10.3 | 9.6 | 11.1 |
| | Group B | Pre-BST | 273 | 263 | 96.3 | 93.4 | 98.2 | 62 | 22.7 | 17.9 | 28.1 | 12.2 | 11.3 | 13.1 |
| | Control | Pre-BST | 280 | 260 | 92.9 | 89.2 | 95.6 | 43 | 15.4 | 11.3 | 20.1 | 10.4 | 9.6 | 11.2 |

Group A = Subjects who received DTPa-IPV/Hib vaccine at 2, 3, 4 months of age in the primary study

Group B = Subjects who received DTPa-IPV/Hib vaccine at 3, 4, 5 months of age in the primary study

Control = Subjects who received DTPa/Hib + IPV vaccines at 2, 3, 4 months of age in the primary study

Seropositivity =Anti-PT antibody concentration ≥ 5 ELU/ml

GMC = geometric mean antibody concentration calculated on all subjects

N = number of subjects with available results

n/% = number/percentage of subjects with concentration equal to or above specified value

95% CI = 95% confidence interval; LL = Lower Limit, UL = Upper Limit

Pre-BST=Pre-booster vaccination blood sampling time point

Template 14 Seroprotection rates and geometric mean titres (GMT) for anti-Poliovirus 1, 2 and 3 antibody by groups at pre vaccination (ATP cohort for analysis of antibody persistence)

| | | | | | ≥ 8 ED <sub>50</sub> | | | | GMT | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | 95% CI | | | 95% CI | |
| Antibody | Group | Timing | N | n | % | LL | UL | value | LL | UL |
| Anti-Poliovirus 1 | Group A | Pre-BST | 272 | 259 | 95.2 | 92.0 | 97.4 | 72.3 | 62.4 | 83.7 |
| | Group B | Pre-BST | 273 | 267 | 97.8 | 95.3 | 99.2 | 95.7 | 82.5 | 111.0 |
| | Control | Pre-BST | 280 | 270 | 96.4 | 93.5 | 98.3 | 77.2 | 67.0 | 89.0 |
| Anti-Poliovirus 2 | Group A | Pre-BST | 272 | 248 | 91.2 | 87.2 | 94.3 | 57.3 | 47.0 | 70.0 |
| | Group B | Pre-BST | 273 | 261 | 95.6 | 92.4 | 97.7 | 63.6 | 53.5 | 75.5 |
| | Control | Pre-BST | 280 | 250 | 89.3 | 85.1 | 92.7 | 42.6 | 35.7 | 50.8 |
| Anti-Poliovirus 3 | Group A | Pre-BST | 272 | 254 | 93.4 | 89.7 | 96.0 | 71.3 | 60.1 | 84.7 |
| | Group B | Pre-BST | 273 | 259 | 94.9 | 91.5 | 97.2 | 79.9 | 66.4 | 96.2 |
| | Control | Pre-BST | 280 | 257 | 91.8 | 87.9 | 94.7 | 60.6 | 51.2 | 71.8 |

Group A = Subjects who received DTPa-IPV/Hib vaccine at 2, 3, 4 months of age in the primary study

Group B = Subjects who received DTPa-IPV/Hib vaccine at 3, 4, 5 months of age in the primary study

Control = Subjects who received DTPa/Hib + IPV vaccines at 2, 3, 4 months of age in the primary study

Seroprotection=Anti-Poliovirus 1, 2 and 3 antibodies ≥8 ED<sub>50</sub>

GMT = geometric mean antibody titre calculated on all subjects

N = number of subjects with available results

n/% = number/percentage of subjects with titre equal to or above specified value

95% CI = 95% confidence interval; LL = Lower Limit, UL = Upper Limit

Pre-BST=Pre-booster vaccination blood sampling time point

Template 15 Difference between groups in percentage of subjects with titre/concentrations equal to or above the proposed cut-off one month after primary vaccination between Form A and Control groups - Inferential analysis (ATP cohort for immunogenicity)

| | Threshold (unit) | | | | | | | Difference in percentage (Control minus FormA) | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Control | | | FormA | | | | 95% CI | |
| Antibody | | N | n | % | N | n | % | % | LL | UL |
| Anti-D | 0.1 IÚ/mL | 219 | 219 | 100 | 214 | 214 | 100 | 0.00 | -2.25 | 2.30 |
| Anti-T | 0.1 IU/mL | 219 | 219 | 100 | 214 | 214 | 100 | 0.00 | -2.25 | 2.30 |
| Polio 1 | 8 | 219 | 219 | 100 | 214 | 214 | 100 | 0.00 | -2.25 | 2.30 |
| Polio 2 | 8 | 219 | 219 | 100 | 214 | 214 | 100 | 0.00 | -2.25 | 2.30 |
| Polio 3 | 8 | 219 | 219 | 100 | 214 | 214 | 100 | 0.00 | -2.25 | 2.30 |
| PT | 10 IU/mL | 219 | 219 | 100 | 214 | 214 | 100 | 0.00 | -2.25 | 2.30 |
| FHA | 10 IU/mL | 219 | 219 | 100 | 214 | 214 | 100 | 0.00 | -2.25 | 2.30 |

FormA = DTPa-HBV-IPV/Hib Form A + Prevenar 13 at 2, 3 and 4 months of age Control = DTPa-HBV-IPV/Hib licensed + Prevenar 13 at 2, 3 and 4 months of age

n/% = number/percentage of subjects with concentration and titre within the specified range 97.5% CI = Standardized asymptotic 97.5% confidence interval; LL = lower limit, UL = upper limit

N = number of subjects with available results
Template 16 Reverse Cumulative curves for anti-rotavirus IgA antibody concentrations at Visit 3 from a subset of subjects - ATP cohort for immunogenicity



### Template 17 Number and percentage of subjects who received study vaccine doses by vaccine (Total vaccinated cohort)

| | Н | paHAV<br>AVRIX<br>I = 182 | dTpa<br>dT <sub>l</sub><br>N = | oa | НА | VdTpa<br>.VRIX<br>= 139 | d | VdTpa<br>Tpa<br>= 139 |
|---|---|---|---|---|---|---|---|---|
| Total number of doses received | n | % | n | % | n | % | n | % |
| 0 | 0 | 0.0 | 1 | 0.5 | 0 | 0.0 | 1 | 0.7 |
| 1 | 182 | 100 | 181 | 99.5 | 139 | 100 | 138 | 99.3 |
| Any | 182 | 100 | 181 | 99.5 | 139 | 100 | 138 | 99.3 |

dTpaHAV = #1 dTpa vaccine(D37750B2)#2 HAV vaccine(DVHA821D2)

HAVdTpa = #1 HAV vaccine(DVHA821D2)#2 dTpa vaccine(D37750B2)

N = number of subjects in each group included in the considered cohort

n/% = number/percentage of subjects receiving the specified total number of doses

Any = number and percentage of subjects receiving at least one dose

Data source = Appendix table IG

#### **Template 18 Compliance in returning symptom sheets (Total vaccinated cohort)**

| Dose | Group | Number<br>of<br>doses | Doses<br>NOT<br>according to<br>protocol | Number<br>of<br>general SS | Compliance<br>%<br>general SS |
|---|---|---|---|---|---|
| 1 | HRV | 508 | 0 | 508 | 100 |
| | Placebo | 257 | 0 | 257 | 100 |
| 2 | HRV | 499 | 0 | 499 | 100 |
| | Placebo | 250 | 0 | 250 | 100 |
| Total | HRV | 1007 | 0 | 1007 | 100 |
| | Placebo | 507 | 0 | 507 | 100 |

SS = Symptom sheets used for the collection of general solicited AEs

Compliance % = (number of doses with symptom sheet return / number of administered doses) X 100

### Template 19 Incidence and nature of symptoms (solicited and unsolicited) reported during the 8-day (Days 0-7) post-vaccination period following each dose and overall (Total vaccinated cohort)

| | | Α | ny | sy | mp | tom | Ge | ne | ral s | symp | toms | Lc | са | l sy | mpt | oms |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95% | <b>6 CI</b> | | | | 959 | % CI | | | | 95% | <b>6 CI</b> |
| | Group | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| Dose 1 | HPV_2D | | | | | | | | | | | | | | | |
| | MMR_DTPa | | | | | | | | | | | | | | | |
| Dose 2 | HPV_2D | | | | | | | | | | | | | | | |
| | MMR_DTPa | | | | | | | | | | | | | | | |
| Overall/dose | HPV_2D | | | | | | | | | | | | | | | |
| | MMR_DTPa | | | | | | | | | | | | | | | |
| Overall/subj | HPV_2D | | | | | | | | | | | | | | | |
| | MMR DTPa | | | | | | | | | | | | | | | |

HPV\_2D = females aged 4-6 years who received two doses of HPV-16/18 L1 VLP AS04 vaccine at Day 0 and Month 6 MMR\_DTPa = females aged 4-6 years who received MMR vaccine at Day 0 and DTPa vaccine at Month 6 For each dose and overall/subject:

N= number of subjects with at least one administered dose

n/%= number/percentage of subjects presenting at least one type of symptom

For overall/dose:

N= number of administered doses

n/%= number/percentage of doses followed by at least one type of symptom

95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

Template 20 Incidence of solicited local symptoms reported during the 7-day (Days 0-6) post-vaccination period following each dose and overall (Total vaccinated cohort)

| | | HPV_2D | | | | | I | MI | ИR | R_DTPa | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 95 % CI | | | | | | 95 | % CI | | |
| Symptom | Туре | N | n | % | LL | UL | N | n | % | LL | UL |
| Pain | All | | | | | | | | | | |
| | Grade 3 | | | | | | | | | | |
| | Medical advice | | | | | | | | | | |
| Redness (mm) | All | | | | | | | | | | |
| , , | >20 | | | | | | | | | | |
| | Medical advice | | | | | | | | | | |
| Swelling (mm) | All | | | | | | | | | | |
| | >20 | | | | | | | | | | |
| | Medical advice | | | | | | | | | | |

HPV\_2D = females aged 4-6 years who received two doses of HPV-16/18 L1 VLP AS04 vaccine at Day 0 and Month 6 MMR\_DTPa = females aged 4-6 years who received MMR vaccine at Day 0 and DTPa vaccine at Month 6

N = number of subjects with an administered dose

n/% = number/percentage of subjects reporting the symptom at least once

# Template 21 Incidence of solicited general symptoms reported during the 7-day (Days 0-6) post-vaccination period following each dose and overall (Total vaccinated cohort)

| | | HPV_2D<br>95 % C | | | | | ΜN | IR | _DT | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | % C |
| Symptom | Type | Nn | % | LL | UL | N | n | % | LL | UL |
| | Dose 1 | | | | • | • | | | , | |
| Each symptom except fever | All | | | | | | | | | |
| | Grade 3 | | | | | | | | | |
| | Related | | | | | | | | | |
| | Grade 3 Related | | | | | | | | | |
| | Medical advice | | | | | | | | | |
| Fever/(Axillary) (°C) | All | | | | | | | | | |
| r even(r willary) ( 'O') | ≥37.5 | | | | | | | | | |
| | >38.0 | | | | | | | | | |
| | >38.5 | | | | | | | | | |
| | >39.0 | | | | | | | | | |
| | >39.5 | | | | | | | | | |
| | >40.0 | | | | | | | | | |
| | Related | | | | | | | | | |
| | >38.0 Related | | | | | | | | | |
| | >38.5 Related | | | | | | | | | |
| | >39.0 Related | | | | | | | | | |
| | >39.5 Related | | | | | | | | | |
| | >40.0 Related | | | | | | | | | |
| | Medical advice | | | | | | | | | |
| | Dose 2 | | 1 | l . | | - | 11 | | l | 1 |
| Each symptom except fever | All | | | | | | | | | |
| | Grade 3 | | | | | | | | | |
| | Related | | | | | | | | | |
| | Grade 3 Related | | | | | | | | | |
| | Medical advice | | | | | | | | | |
| Fever/(Axillary) (°C) | All | | | | | | | | | |
| rever/(Axillary) ( C) | ≥37.5 | | | | | | | | | |
| | >38.0 | | | | | | | | | |
| | >38.5 | | | | | | | | | |
| | >39.0 | | | | | | | | | |
| | >39.5 | | | | | | | | | |
| | >40.0 | | | | | | | | | |
| | Related | | | | | | | | | |
| | >38.0 Related | | | | | | | | | |
| | >38.5 Related | | | | | | | | | |
| | >39.0 Related | | | | | | | | | |
| | >39.5 Related | | | | | | | | | |
| | >40.0 Related | | | | | | | | | |
| | Medical advice | | | | | | | | | |
| | Overall/dose | 1 1 | | | 1 | <u> </u> | ı | | | - |
| Each symptom except fever | All | | | | | | | | | |
| symptom ondoperotor | Grade 3 | | | | | H | H | | | |
| | Related | | | | 1 | | | | | |
| | Grade 3 Related | + | | | | | | | | |
| | Medical advice | | | | | | $\vdash$ | | | |
| Fover//Avilland (90) | All | | | | | | | | | |
| Fever/(Axillary) (°C) | | | | | | - | Н | | | |
| | ≥37.5 | | | | | | | | | |
| | >38.0 | | | | | | | | | |

114720 (ROTA-079) Statistical Analysis Plan

| | | HPV_2D<br>95 % CI | | | | | MI | ИR | _DT | Ра | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | 95 ° | % C | | |
| Symptom | Туре | N | n | % | LL | UL | N | n | % | LL | UL |
| | >38.5 | | | | | | | | | | |
| | >39.0 | | | | | | | | | | |
| | >39.5 | | | | | | | | | | |
| | >40.0 | | | | | | | | | | |
| | Related | | | | | | | | | | |
| | >38.0 Related | | | | | | | | | | |
| | >38.5 Related | | | | | | | | | | |
| | >39.0 Related | | | | | | | | | | |
| | >39.5 Related | | | | | | | | | | |
| | >40.0 Related | | | | | | | | | | |
| | Medical advice | | | | | | | | | | |
| | Overall/subject | | | | | | | | | | |
| Each symptom except fever | All | | | | | | | | | | |
| | Grade 3 | | | | | | | | | | |
| | Related | | | | | | | | | | |
| | Grade 3 Related | | | | | | | | | | |
| | Medical advice | | | | | | | | | | |
| Fever/(Axillary) (°C) | All | | | | | | | | | | |
| , ,,,, | ≥37.5 | | | | | | | | | | |
| | >38.0 | | | | | | | | | | |
| | >38.5 | | | | | | | | | | |
| | >39.0 | | | | | | | | | | |
| | >39.5 | | | | | | | | | | |
| | >40.0 | | | | | | | | | | |
| | Related | | | | | | | | | | |
| | >38.0 Related | | | | | | | | | | |
| | >38.5 Related | | | | | | | | | | |
| | >39.0 Related | | | | | | | | | | |
| | >39.5 Related | | | | | | | | | | |
| | >40.0 Related | | | | | | | | | | |
| | Medical advice | | | | | | | | | | |

HPV\_2D = females aged 4-6 years who received two doses of HPV-16/18 L1 VLP AS04 vaccine at Day 0 and Month 6 MMR\_DTPa = females aged 4-6 years who received MMR vaccine at Day 0 and DTPa vaccine at Month 6 For each dose and overall/subject:

N = number of subjects with at least one administered dose

n/% = number/percentage of subjects reporting the symptom at least once For Overall/dose:

N = number of administered doses

n/% = number/percentage of doses followed by at least one type of symptom

114720 (ROTA-079) Statistical Analysis Plan

## Template 22 Incidence of solicited local symptoms reported during the 7-day (Days 0-6) post-vaccination period following each dose and overall (Total vaccinated cohort)

| | | HPV_2D | | | | | I | MI | ИR | _DT | Ра |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 95 % CI | | | % CI | | | | 95 | % CI | |
| Symptom | Туре | N | n | % | LL | UL | N | n | % | LL | UL |
| Pain | All | | | | | | | | | | |
| | Grade 3 | | | | | | | | | | |
| | Medical advice | | | | | | | | | | |
| Redness (mm) | All | | | | | | | | | | |
| , , | >20 | | | | | | | | | | |
| | Medical advice | | | | | | | | | | |
| Swelling (mm) | All | | | | | | | | | | |
| | >20 | | | | | | | | | | |
| | Medical advice | | | | | | | | | | |

HPV\_2D = females aged 4-6 years who received two doses of HPV-16/18 L1 VLP AS04 vaccine at Day 0 and Month 6 MMR\_DTPa = females aged 4-6 years who received MMR vaccine at Day 0 and DTPa vaccine at Month 6 N = number of subjects with a documented dose

n/% = number/percentage of subjects reporting the symptom at least once 95%CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

## Template 23 Incidence of solicited general symptoms reported during the 7-day (Days 0-6) post-vaccination period following each dose and overall (Total vaccinated cohort)

| | | HPV_2D | | | | | | M۱ | ΙR | _D1 | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 95 % C<br>N n % LL UL | | | | | | | | | % CI |
| Symptom | Type | N | n | % | LL | UL | N | n | % | LL | UL |
| | Dose 1 | | | | ı | | | | | | |
| Each symptom except fever | All | | | | | | | | | | |
| | Grade 3 | | | | | | | | | | |
| | Related | | | | | | | | | | |
| | Grade 3 Related | | | | | | | | | | |
| | Medical advice | | | | | | | | | | |
| Fever/(Axillary) (°C) | All | | | | | | | | | | |
| | ≥37.5 | | | | | | | | | | |
| | >38.0 | | | | | | | | | | |
| | >38.5 | | | | | | | | | | |
| | >39.0 | | | | | | | | | | |
| | >39.5 | | | | | | | | | | |
| | >40.0 | | | | | | | | | | |
| | Related | | | | | | | | | | |
| | >38.0 Related | | | | | | | | | | |
| | >38.5 Related | | | | | | | | | | |
| | >39.0 Related | | | | | | | | | | |
| | >39.5 Related | | | | | | | | | | |
| | >40.0 Related | | | | | | | | | | |
| | Medical advice | | | | | | | | | | |
| | Dose 2 | | | | | 1 | | | | | 1 |
| Each symptom except fever | All | | | | | | | | | | |
| , , | Grade 3 | | | | | | | | | | |
| | Related | | | | | | | | | | |
| | Grade 3 Related | | | | | | | | | | |
| | Medical advice | | | | | | | | | | |
| Fever/(Axillary) (°C) | All | | | | | | | | | | |
| ( 7) ( ) | ≥37.5 | | | | | | | | | | |
| | >38.0 | | | | | | | | | | |
| | >38.5 | | | | | | | | | | |
| | >39.0 | | | | | | | | | | |
| | >39.5 | | | | | | | | | | |
| | >40.0 | | | | | | | | | | |
| | Related | | | | | | | | | | |
| | >38.0 Related | | | | | | | | | | |
| | >38.5 Related | | | | | | | | | | |
| | >39.0 Related | | | | | | | | | | |
| | >39.5 Related | | | | | | | | | | |
| | >40.0 Related | | | | | | | | | | |
| | Medical advice | | | | | | | | | | |
| | Overall/dose | 1 | | | | 1 | | | | | |
| Each symptom except fever | All | | Τ | | | | | | | | 1 |
| Lacit symptom except level | Grade 3 | | | | | | | | | | |
| | Related | 1 | | | | | | | | | |
| | Grade 3 Related | H | $\vdash$ | | | | | | | | |
| | Medical advice | - | $\vdash$ | | | | | - | | | |
| Eover//Avillan/\ /°C\ | All | - | $\vdash$ | | | 1 | | | | | |
| Fever/(Axillary) (°C) | | | $\vdash$ | | | 1 | | | | | |
| | ≥37.5 | _ | - | | | 1 | | - | | | |
| | >38.0 | | | | | | | | | | |

114720 (ROTA-079) Statistical Analysis Plan

| | | HPV_2D<br>95 % C | | | | | MI | ۷R | _DT | Ра | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 95 % C<br>N n % LL UL | | | % CI | | | | 95 | % CI | |
| Symptom | Туре | N | n | % | LL | UL | N | n | % | LL | UL |
| | >38.5 | | | | | | | | | | |
| | >39.0 | | | | | | | | | | |
| | >39.5 | | | | | | | | | | |
| | >40.0 | | | | | | | | | | |
| | Related | | | | | | | | | | |
| | >38.0 Related | | | | | | | | | | |
| | >38.5 Related | | | | | | | | | | |
| | >39.0 Related | | | | | | | | | | |
| | >39.5 Related | | | | | | | | | | |
| | >40.0 Related | | | | | | | | | | |
| | Medical advice | | | | | | | | | | |
| | Overall/subject | | | | | 1 | | | ! | | J |
| Each symptom except fever | All | | | | | | | | | | |
| , | Grade 3 | | | | | | | | | | |
| | Related | | | | | | | | | | |
| | Grade 3 Related | | | | | | | | | | |
| | Medical advice | | | | | | | | | | |
| Fever/(Axillary) (°C) | All | | | | | | | | | | |
| | ≥37.5 | | | | | | | | | | |
| | >38.0 | | | | | | | | | | |
| | >38.5 | | | | | | | | | | |
| | >39.0 | | | | | | | | | | |
| | >39.5 | | | | | | | | | | |
| | >40.0 | | | | | | | | | | |
| | Related | | | | | | | | | | |
| | >38.0 Related | | | | | | | | | | |
| | >38.5 Related | | | | | | | | | | |
| | >39.0 Related | | | | | | | | | | |
| | >39.5 Related | | | | | | | | | | |
| | >40.0 Related | | | | | | | | | | |
| | Medical advice | | | | | | | | | | |

N = number of subjects with at least one documented dose

n/% = number/percentage of subjects reporting the symptom at least once

For Overall/dose:

N = number of documented doses

n/% = number/percentage of doses followed by at least one type of symptom

114720 (ROTA-079) Statistical Analysis Plan

# Template 24 Percentage of subjects reporting the occurrence of unsolicited symptoms classified by MedDRA Primary System Organ Class within the 31-day (Days 0-30) post-vaccination period (Total vaccinated cohort)

| | | | HF | PV_2<br>N = | | M | | _DT<br>N = | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | 6 CI | | | | % CI |
| Primary System Organ Class (CODE) | Preferred Term (CODE) | n | % | LL | UL | n | % | LL | UL |
| At least one symptom | | | | | | | | | |
| Blood and lymphatic system disorders (10005329) | Anaemia (10002034) | | | | | | | | |
| Ear and labyrinth disorders (10013993) | Ear pain (10014020) | | | | | | | | |
| Gastrointestinal disorders (10017947) | Abdominal pain (10000081) | | | | | | | | |
| | Abdominal pain upper (10000087) | | | | | | | | |
| | Anal fissure (10002153) | | | | | | | | |

HPV\_2D = females aged 4-6 years who received two doses of HPV-16/18 L1 VLP AS04 vaccine at Day 0 and Month 6 MMR\_DTPa = females aged 4-6 years who received MMR vaccine at Day 0 and DTPa vaccine at Month 6 At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with at least one administered dose

n/% = number/percentage of subjects reporting the symptom at least once

n/% = number/percentage of subjects reporting the symptom at least once 95% CI = exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

## Template 25 Percentage of doses with unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term within the 43-day (Days 0-42) post-vaccination period (Total vaccinated cohort)

| | | | HF | PV_2<br>N = | | M | | _D1<br>N = | ГРа |
|---|---|---|---|---|---|---|---|---|---|
| | | | | 95% | 6 CI | | | 95% | <b>6 CI</b> |
| Primary System Organ Class (CODE) | Preferred Term (CODE) | n | % | LL | UL | n | % | LL | UL |
| At least one symptom | | | | | | | | | |
| Blood and lymphatic system disorders (10005329) | Anaemia (10002034) | | | | | | | | |
| Ear and labyrinth disorders (10013993) | Ear pain (10014020) | | | | | | | | |
| Gastrointestinal disorders (10017947) | Abdominal pain (10000081) | | | | | | | | |
| , , | Abdominal pain upper (10000087) | | | | | | | | |
| | Anal fissure (10002153) | | | | | | | | |

HPV\_2D = females aged 4-6 years who received two doses of HPV-16/18 L1 VLP AS04 vaccine at Day 0 and Month 6 MMR\_DTPa = females aged 4-6 years who received MMR vaccine at Day 0 and DTPa vaccine at Month 6 At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term) N = number of administered doses

n (%) = number (percentage) of doses with the symptom

114720 (ROTA-079) Statistical Analysis Plan

### Template 26 Listing of dropouts due to AEs, SAEs and solicited symptoms (Total cohort)

| Study-<br>Subject<br>No. | Country | Gender | AE Description | SAE | Causality | Outcome | Type of discontinuation |
|---|---|---|---|---|---|---|---|
| PP<br>D | Germany | F | SUBJECT DIED | Υ | | Fatal | Study at visit/contact: VISIT11 (Y5) |
| D D | Germany | F | SUBJECT DIED | Υ | | Fatal | Study at visit/contact: VISIT11 (Y5) |

114720 (ROTA-079) Statistical Analysis Plan

### Template 27 Listings of SAEs (Total vaccinated cohort)

| Sub. | Case Id | Age at | Sex | Verbatim | Preferred | System Organ Class | MA | Dose | Day of | Durati | Intensity | Causality | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| No. | | onset | | | term | | type | | onset | on | | | |
| | | (Week) | | | | | | | | | | | |
| P | PPD | 37 | F | Blinded | Blinded | Infections and infestations | НО | 2 | 177 | 6 | 2 | N | Recovered/resolved |
| Р | PPD | 38 | F | Blinded | Blinded | Infections and infestations | НО | 2 | 182 | 10 | 2 | N | Recovered/resolved |
| | PPD | 66 | F | Blinded | Blinded | Respiratory, thoracic and mediastinal disorders | НО | 2 | 375 | 7 | 2 | N | Recovered/resolved |
| | | 66 | | Blinded | Blinded | Infections and infestations | НО | 2 | 375 | 5 | 2 | N | Recovered/resolved |
| Р | PPD | 78 | M | Blinded | Blinded | Infections and infestations | НО | 2 | 467 | 8 | 2 | N | Recovered/resolved |
| P | PPD | 56 | F | Blinded | Blinded | Infections and infestations | НО | 2 | 299 | 13 | 2 | N | Recovered/resolved |
| Р | | 56 | | Blinded | Blinded | Blood and lymphatic system disorders | НО | 2 | 299 | 133 | 2 | N | Recovered/resolved |
| | PPD | 59 | F | Blinded | Blinded | Infections and infestations | НО | 2 | 319 | 11 | 2 | N | Recovered/resolved |
| | PPD | 73 | F | Blinded | Blinded | Infections and infestations | ER | 2 | 417 | 5 | 2 | N | Recovered/resolved |
| PP | PPD | 13 | М | Blinded | Blinded | Infections and infestations | НО | 2 | 15 | 17 | 1 | N | Recovered/resolved |
| D | | 13 | | Blinded | Blinded | Infections and infestations | НО | 2 | 17 | 8 | 2 | N | Recovered/resolved |
| PP | PPD | 25 | М | Blinded | Blinded | Infections and infestations | НО | 2 | 90 | 15 | 2 | N | Recovered/resolved |
| PP<br>D | PPD | 24 | М | Blinded | Blinded | Musculoskeletal and connective tissue disorders | НО | 2 | 76 | 31 | 1 | N | Recovered/resolved |

HO = hospitalisation

MD = Medical Personnel

12-SEP-2016 Page 47 of 51

## Template 28 Number and percentage of doses and of subjects who took at least one concomitant medication during the study period (from Dose 1 till database lock) by type (Total vaccinated cohort)

| | HRV | | | | Placebo | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 95% | 6 CI | | | | 959 | % CI |
| | N | n | % | LL | UL | N | n | % | LL | UL |
| Dose 1 | | | | | | | | | | |
| Any | 508 | 165 | 32.5 | 28.4 | 36.7 | 257 | 70 | 27.2 | 21.9 | 33.1 |
| Any antipyretic | 508 | 16 | 3.1 | 1.8 | 5.1 | 257 | 13 | 5.1 | 2.7 | 8.5 |
| Prophylactic antipyretic | 508 | 0 | 0.0 | 0.0 | 0.7 | 257 | 0 | 0.0 | 0.0 | 1.4 |
| Any antibiotic | 508 | 59 | 11.6 | 9.0 | 14.7 | 257 | 22 | 8.6 | 5.4 | 12.7 |
| Dose 2 | | | | | | | | | | |
| Any | 499 | 217 | 43.5 | 39.1 | 48.0 | 250 | 122 | 48.8 | 42.5 | 55.2 |
| Any antipyretic | 499 | 32 | 6.4 | 4.4 | 8.9 | 250 | 21 | 8.4 | 5.3 | 12.6 |
| Prophylactic antipyretic | 499 | 0 | 0.0 | 0.0 | 0.7 | 250 | 0 | 0.0 | 0.0 | 1.5 |
| Any antibiotic | 499 | 105 | 21.0 | 17.5 | 24.9 | 250 | 51 | 20.4 | 15.6 | 25.9 |
| | | • | Overal | I/dose | | | | | | |
| Any | 1007 | 382 | 37.9 | 34.9 | 41.0 | 507 | 192 | 37.9 | 33.6 | 42.3 |
| Any antipyretic | 1007 | 48 | 4.8 | 3.5 | 6.3 | 507 | 34 | 6.7 | 4.7 | 9.2 |
| Prophylactic antipyretic | 1007 | 0 | 0.0 | 0.0 | 0.4 | 507 | 0 | 0.0 | 0.0 | 0.7 |
| Any antibiotic | 1007 | 164 | 16.3 | 14.1 | 18.7 | 507 | 73 | 14.4 | 11.5 | 17.8 |
| Overall/subject | | | | | | | | | | |
| Any | 508 | 300 | 59.1 | 54.6 | 63.4 | 257 | 155 | 60.3 | 54.0 | 66.3 |
| Any antipyretic | 508 | 43 | 8.5 | 6.2 | 11.2 | 257 | 32 | 12.5 | 8.7 | 17.1 |
| Prophylactic antipyretic | 508 | 0 | 0.0 | 0.0 | 0.7 | 257 | 0 | 0.0 | 0.0 | 1.4 |
| Any antibiotic | 508 | 152 | 29.9 | 26.0 | 34.1 | 257 | 65 | 25.3 | 20.1 | 31.1 |

For each dose and overall/subject:

For overall/dose:

N= number of administered doses

n (%)= number (percentage) of doses after which the specified concomitant medication was started at least once during the mentioned period

95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

Database lock date = 31 Mar 2009

N= number of subjects with at least one administered dose

n (%)= number (percentage) of subjects who started to take the specified concomitant medication at least once during the mentioned period

## Template 29 Incidence of solicited general symptoms reported during the 7-day (Days 0-6) post-vaccination period following each dose and overall (Total vaccinated cohort)

| | | | HPV | | | V_2D | | | ИR | _DT | Ра |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | % CI | | | | | % CI |
| Symptom | Туре | N | n | % | LL | UL | N | n | % | LL | UL |
| | Dose 1 | | | | | | | | | • | |
| Each symptom except fever | All | | | | | | | | | | |
| | Grade 3 | | | | | | | | | | |
| | Related | | | | | | | | | | |
| Fever/(Axillary) (°C) | All | | | | | | | | | | |
| | >39.0 | | | | | | | | | | |
| | Related | | | | | | | | | | |
| | Dose 2 | | | | | | | | | | |
| Each symptom except fever | All | | | | | | | | | | |
| | Grade 3 | | | | | | | | | | |
| | Related | | | | | | | | | | |
| Fever/(Axillary) (°C) | All | | | | | | | | | | |
| , ,,,, | >39.0 | | | | | | | | | | |
| | Related | | | | | | | | | | |
| | Dose 3 | | | | | | | | | | |
| Each symptom except fever | All | | | | | | | | | | |
| | Grade 3 | | | | | | | | | | |
| | Related | | | | | | | | | | |
| Fever/(Axillary) (°C) | All | | | | | | | | | | |
| | >39.0 | | | | | | | | | | |
| | Related | | | | | | | | | | |
| | Across Dos | es | | | | | | | | | |
| Each symptom except fever | All | | | | | | | | | | |
| , , , , | Grade 3 | | | | | | | | | | |
| | Related | | | | | | | | | | |
| Fever/(Axillary) (°C) | All | | | | | | | | | | |
| | >39.0 | | | | | | | | | | |
| | Related | | | | | | | | | | |

HPV\_2D = females aged 4-6 years who received two doses of HPV-16/18 L1 VLP AS04 vaccine at Day 0 and Month 6 MMR\_DTPa = females aged 4-6 years who received MMR vaccine at Day 0 and DTPa vaccine at Month 6 N = number of subjects with at least one administered dose

n/% = number/percentage of subjects reporting the symptom at least once

### Template 30 Number (%) of subjects with serious adverse events from first study vaccination up to Visit 7 including number of events reported (Total vaccinated cohort)

| | | | Gr 1<br>N = | | | | Gr2<br>N = | |
|---|---|---|---|---|---|---|---|---|
| Type of Event | Primary System Organ<br>Class | Preferred Term<br>(CODE) | n* | n | % | n* | n | % |
| SAE | At least one symptom | | | | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | | | | |
| Related SAE | At least one symptom | | | | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | | | | |
| Fatal SAE | At least one symptom | | | | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | | | | |
| Related fatal SAE | At least one symptom | | | | | | | |
| | <each soc=""></each> | <each pt="" term=""></each> | | | | | | |

Gr 1 = Group 1 description

Template 31 Solicited and unsolicited symptoms experienced by at least 5 % of subjects classified by MedDRA Primary System Organ Class and Preferred Term within 31-day (Days 0-30) post-vaccination period after any dose of liquid HRV vaccine and first dose of DPT-IPV vaccine - SAE excluded (Total vaccinated cohort)

| | | Н | IPV_<br>N : | | MMF | R_D<br>N = | |
|---|---|---|---|---|---|---|---|
| Primary System Organ Class (CODE) | Preferred Term (CODE) | n* | n | % | n* | n | % |
| At least one symptom | | | | | | | |
| <each soc=""></each> | <each pt="" term=""></each> | | | | | | |

HPV\_2D = females aged 4-6 years who received two doses of HPV-16/18 L1 VLP AS04 vaccine at Day 0 and Month 6 MMR\_DTPa = females aged 4-6 years who received MMR vaccine at Day 0 and DTPa vaccine at Month 6 At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with the administered dose

n/% = number/percentage of subjects reporting the symptom at least once

Gr 2 = Group 2 description

N = number of subjects with the administered dose

n\* = number of events reported

n/% = number/percentage of subjects reporting the symptom at least once

n\* = number of events reported

114720 (ROTA-079) Statistical Analysis Plan

### Template 32 Number of enrolled subjects by age category (Total vaccinated cohort)

| | | Gr 1<br>N = | Gr 2<br>N = | Gr 3<br>N = | Total<br>N = |
|---|---|---|---|---|---|
| Characteristics | Categories | n | n | n | n |
| Age category | In utero | | | | |
| | Preterm newborn infants<br>(gestational age < 37 wks)<br>Newborns (0-27 days) | | | | |
| | Infants and toddlers (28 days-<br>23 months) | | | | |
| | Children (2-11 years) | | | | |
| | Adolescents (12-17 years) | | | | |
| | Adults (18-64 years) | | | | |
| | From 65-84 years | | | | |
| | 85 years and over | | | | |
| | Missing | | | | |

Gr 1 = Group 1 description

n= number of enrolled subjects included in each group or in total for a given age category or for all age categories Missing = <describe missing>

Gr 2 = Group 2 description

Gr 3 = Group 3 description

N = Number of enrolled subjects